CLINICAL TRIAL: NCT07213258
Title: CHAMPION: Combining HIV And Meth Prevention and Treatment Interventions Optimized for HIV-Negative MSM
Acronym: CHAMPION
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Kiyomi Tsuyuki, Multi-Principal Investigator, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R21DA060856 (NIH); R21DA060856 (NIH)
Record Dates: First submitted 2025-01-24; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: PrEP Adherence; Methamphetamine Use Disorder; HIV
Keywords: MSM; HIV Negative; mild MUD; moderate MUD; Methamphetamine Use Disorder (MUD); CBT4CBT; PrEPAPP; mHealth; Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CHAMPION Intervention Arm (Experimental): mHealth app to track and promote PrEP adherence using motivational messages combined with computer-administered cognitive behavioral therapy for the full 6-month period.
  Interventions: Behavioral: CHAMPION Intervention
- Waitlist Control Arm (Other): 3-month waitlist period including informational resources, followed by 3-month CHAMPION intervention.
  Interventions: Behavioral: Delayed CHAMPION Package

INTERVENTIONS:
Behavioral: CHAMPION Intervention — MHealth intervention to enhance PrEP adherence, combined with computer-administered cognitive behavioral therapy for a 6-month period for the intervention arm.
  Arms: CHAMPION Intervention Arm
Behavioral: Delayed CHAMPION Package — Informational resources for first 3-months of study, followed by CHAMPION intervention for final 3-months.
  Arms: Waitlist Control Arm

SUMMARY:
The goal of this randomized controlled trial is to pilot test new mobile health (mHealth) interventions to improve PrEP adherence among HIV-negative men who have sex with men (MSM) with mild to moderate methamphetamine use disorder (MUD). The CHAMPION intervention combines two mHealth tools-PrEPAPP and CBT4CBT-to address both HIV prevention and MUD treatment needs in this population. The study's specific aims are:

* To evaluate the feasibility and acceptability of the CHAMPION intervention based on treatment retention and engagement rates.
* To examine the preliminary efficacy the CHAMPION intervention to improve PrEP adherence, as measured by dried blood spot (DBS) tests compared to the waitlist control group.

DETAILED DESCRIPTION:
The CHAMPION (Combining HIV And Meth Prevention and Treatment Interventions Optimized for HIV-Negative MSM) study, a randomized controlled trial that aims to pilot test state-of-the-art multi-modal pharmaco-behavioral interventions to increase PrEP adherence among HIV-negative MSM who use meth, versus a waitlist control. The study will enroll 100 HIV-negative MSM with mild or moderate meth use disorder (MUD) and sub-optimal PrEP adherence. The study will follow participants for 6 months. The intervention arm will receive the 6-month mHealth intervention package, CHAMPION, at baseline, while the waitlist control will receive it at month-3 follow-up. Results of this pilot study will determine the viability of combining interventions that reduce meth use and enhance PrEP adherence, informing the direction of future interventions for MSM who use meth.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-negative
2. Cis-gender male
3. Age 18-40 years old
4. Mild or moderate MUD (by DSM-5 SCID criteria)
5. Anal intercourse with one or more male partners in the past 6 months
6. Started daily oral PrEP more than 30 days ago and self-reported not always taking PrEP as prescribed in the past 30 days (consistent with PrEP It! inclusion criteria)
7. Willingness to participate in an mHealth study with a 6-month follow-up
8. Residing in San Diego or San Francisco County

Exclusion Criteria:

1. Residing outside of San Diego or San Francisco County
2. Any condition that, in the principal investigator's judgment interferes with safe study participation or adherence to study procedures
3. Not able/willing to complete virtual/remote visits
4. Not willing to learn to self-collect dried blood spots using a finger stick

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10-22 (Estimated); Primary Completion 2026-08-15 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
Feasibility & Acceptability of CHAMPION | 6 months
  We will calculate the following feasibility and acceptability measures:
  1. study completion rate (mean, standard deviation)
  2. days of PrEPAPP use (mean, standard deviation)
  3. CBT4CBT virtual sessions completed (mean, standard deviation)
PrEP adherence | 6-Months
  We will examine the preliminary efficacy of CHAMPION vs. a waitlist control on increasing PrEP adherence, compared to a waitlist control as determined by dried blood spot (DBS) tests. In preparation for a larger efficacy trial, we will explore the preliminary efficacy of CHAMPION vs. waitlist control in increasing PrEP adherence. PrEP drug levels in DBS samples will be dichotomized as PrEP adherence, or not, using established cut-offs for protective levels of PrEP. We will calculate the following outcome measure:
  1.) Number and percent adherent to PrEP, based on DBS.

OTHER OUTCOMES:
Meth use | 6 months
  Explored through monthly self-reported data on the CHAMPION App (intervention arm). We will calculate the following outcome:
  1) Days of meth use in the past month (mean, standard deviation)
Sexual risk behavior | 6 months
  To determine the preliminary efficacy in reducing sexual risk behaviors, we will use GEE Poisson, binomial and negative binomial models with robust standard errors to assess evidence that the intervention reduces HIV risk behaviors. We will calculate the following outcomes:
  1. number of sex partners (mean, standard deviation)
  2. number of sex partners with whom meth are used (mean, standard deviation)
  3. episodes of condomless sex with serodiscordant partners (mean, standard deviation)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn-Milo Santos, PhD, MPH, Principal Investigator — University of California, San Francisco; Kiyomi Tsuyuki, PhD, MPH, Principal Investigator — University of California, San Diego
Locations (1):
- Center on Substance Use and Health, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No